CLINICAL TRIAL: NCT05878028
Title: L-TIL Plus Tislelizumab as Second Line Therapy for PD-1 Inhibitor Resistant Advanced NSCLC Patients
Brief Title: L-TIL Plus Tislelizumab for PD1 Antibody Resistant aNSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Quanli Gao (Other Government)
Responsible Party: Sponsor-Investigator, Quanli Gao, Head of Immunotherapy department, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH L-TIL aNSCLC
Record Dates: First submitted 2023-05-06; First posted 2023-05-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: L-TIL; PD1 antibody resistance; Tislizumab; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-TIL plus Tislelizumab and Docetaxel (Experimental): Tislelizumab, 200mg, ivgtt, d1, Q3W for one year L-TIL cells, （3-10）x10^9/m2, ivgtt, d14, Q3W for 4 or 6 cycles Docetacel, 75mg/m2, ivgtt, d1, Q3W for 4 cycles
  Interventions: Combination Product: L-TIL, Tislelizumab, Docetaxel

INTERVENTIONS:
Combination Product: L-TIL, Tislelizumab, Docetaxel — PD1 positive lymphocytes were collect, isolated, and expanded from peripheral blood, then infused back into the patient's body. Besides this, Tislelizumab and Docetaxel were used as combination therapy.
  Other Names: Liquid Tumor Infiltrating Lymphocytes

SUMMARY:
The goal of this observational study is to test in advanced non-small cell lung cancer patients with negative driver gene. For these patients, PD1 antibody therapy combined with chemotherapy was the preferred regimen. However, there is no standard regimen for the patients who refractory from the first-line PD1 inhibitor based therapy.

The main questions they aim to answer are: 1.The efficacy of Liquid Tumor Infiltrating Lymphocytes (L-TIL) plus Tislelizumab and Docetaxel for patients failure from first line chemotherapy and PD1 inhibitor therapy. 2. The safety of L-TIL plus Tislelizumab and Docetaxel as second line therapy.

All participants will receive four cycles of Docetaxel chemotherapy, six cycles of L-TIL cells infusion and one year of Tislelizumab treatment except for disease progression, intolerable toxicity, withdrawal informed consent, death and so on.

DETAILED DESCRIPTION:
This study is one arm, single center, phase II clinical trial. The participants were diagnosed with metastatic non-small cell lung cancer but without actionable biomarkers (eg: EGFR, ALK, MET, ROS1). PD1 inhibitor and chemotherapy as first line therapy was not respond, or develop tumor progression after a response. Four cycles of Docetaxel chemotherapy, six cycles of L-TIL cells infusion and one year of Tislelizumab regimen Q3W were used. Docetacxel was dosed 75mg/m2 and Tislelizumab was dosed 200mg on day 1, L-TIL cells were dosed (3-10)x10*9/m2 on day 14. Eligible patients were no less than 18 and no more than 75 years old, with adequate organ function but without active infection and autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer patients diagnosed by pathological histology.
* Imaging examination showed stage IV disease.
* Non-squamous cancer patients shall be EGFR , ALK, ROS1, RET, MET negative.
* Failure from anti-PD-1 antibody treatment, including treatment ineffective or effective for a period then progress.
* The Eastern Oncology Collaboration Group (ECOG) scores 0-1.
* At least one imaging lesion can be measured, according to the standard for evaluating the effectiveness of solid tumors (RECIST 1.1).
* Asymptomatic or stable symptoms after local treatment is allowed.
* Subjects are allowed to receive palliative radiation.
* Enough organ functions well.
* Patients have good superficial venous blood circulation, which can meet the needs of intravenous dripping.
* No other serious diseases that conflict with this study regimes (e.g. autoimmune diseases, immune deficiencies, organ transplants, chronic infections).
* For female subjects with reproductive age, the pregnancy test should be accepted within 3 days prior to the first study drug administered (day 1 of cycle 1) and the results are negative.
* In the event of a risk of conceival, all subjects (male or female) must adopt contraception at a rate of less than 1% annually for the entire treatment period up to 120 days after the last study of the drug was administered (or 180 days after the last study of the drug).
* The patient himself agrees to participate in this clinical trial, sign the Informed Consent Letter, complete the procedure, treatment, and follow-up.

Exclusion Criteria:

* Small cell lung cancer (SCLC), including mixing pathology, combined with SCLC and NSCLC.
* Accepted radiation treatment in special organ before the first drug was administered, eg: more than 30% bone marrow within 14 days.
* Diagnosed with second malignant diseases within five years.
* Participating in other clinical trial.
* Treatment with other drugs, including thymus peptide, interferon, interleukin, and so on.
* Active autoimmune diseases requires systemic treatment.
* Receiving glucocorticoid therapy, excluding local glucocorticoids in nose, inhalation or other pathways, or any other form of immunosuppressive therapy.
* Uncontrolled chest and abdominal fluid.
* Patients have accepted organ transplantation or hematopoietic stem cell transplantation.
* Allergic to intervention drugs, including ingredients and auxiliary components. ·Incomplete recovery from the adverse events.
* Active hepatitis B or HCV infection.
* Accepted active vaccines within 30 days before the first dose.
* Women who are pregnant or breastfeeding.
* Symptomatic CNS metastasis.
* Uncontrolled active infections, eg. sepsis, mycemia, fungal hematoma.
* With serious mental disorders.
* Other conditions that the researchers believe in having potential risks which are not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 months
  overall response rate (including complete response and partial response)

SECONDARY OUTCOMES:
PFS | 6 months and 12 months
  duration of disease stable or better
DCR | 3 months
  disease control rate (including patients who achieved complete response, partial response and stable disease)
DOR | 6 months and 12 months
  duration of response

CONTACTS AND LOCATIONS:
Overall Officials: YanYan NA Liu, phD, Study Chair — Henan Cancer Hospital
Locations (1):
- No.127 Dongming Road, Zhengzhou, Henan, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT05878028/Prot_SAP_000.pdf